CLINICAL TRIAL: NCT01722617
Title: A Study to Validate Questionnaires FLARE and OM-RA-FLARE Measuring Disease Flares in Patients With Rheumatoid Arthritis.
Acronym: FLARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Régional et Universitaire de Brest (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Grenoble (Other); University Hospital Center of Martinique (Other); University Hospital, Montpellier (Other); Nantes University Hospital (Other); Bichat Hospital (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Poitiers University Hospital (Other); University Hospital, Rouen (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-A01349-32
Record Dates: First submitted 2012-10-26; First posted 2012-11-07 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2012-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DAS 28 (No Intervention): Patients in this group will be asked to fill basic questionnaires, but without the FLARE questionnaires.
- DAS 28 + FLARE questionnaires (Active Comparator): Patients in this group will be asked to fill basic questionnaires and FLARE questionnaires.
  Interventions: Other: Questionnaire
- DAS 28+FLARE + information to doctor (Active Comparator): Patients in this group will fill basic and FLARE questionnaires which then will be transmitted to physician.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients in groups 2 and 3 will be asked to fill in questionnaires FLARE.
  Arms: DAS 28 + FLARE questionnaires; DAS 28+FLARE + information to doctor

SUMMARY:
Rheumatoid arthritis (RA) is a rheumatic inflammatory synovitis characterized by pain and joint swelling as well as thickening synovial (pannus) lesions that are responsible of osteocartilaginous and tendon damage. It evolves in spurts or long and variable intensity interspersed with remissions.

The effectiveness of treatment is based on the proportion of patients who achieve a certain degree of improvement over the initial level of various parameters such as response criteria ACR 20, 50 or 70% or EULAR based on the evolution of DAS 28 or DAS 44. These response criteria are now well validated but do not fully take into account the improvement of the patient's condition. In contrast, there is no questionnaire to identify the proportion of patients whose RA worsened between the medical visits. Such a questionnaire is necessary to detect flares outbreaks in daily practice and in randomized clinical trials, follow-up studies or longitudinal studies after drugs marketing to detect a reversal of disease activity.

Both STPR group and OMERACT group have each developed such a new self-administered questionnaire (FLARE and OM-RA-FLARE) to detect the flare- in RA patients.

The objective of this study is to validate the questionnaires FLARE and OM-RA-FLARE among RA patients using the methodology advocated by the OMERACT in terms of validity (truth), discriminating power (discrimination) and feasibility

DETAILED DESCRIPTION:
There will be 6 months of follow up including 3 medical visits for each patients:

* M0 (medical visit for inclusion)
* follow up between M0 - M3
* M3 (medical visit at 3 months after inclusion)
* follow up between M3 - M6
* M6 (medical visit at 6 months after inclusion)

At the inclusion visit (M0), after the verification of inclusion and non-inclusion criteria, the following information will be collected:

* Socio-demographical data : age, sex, level of education (primary, secondary, college, university), occupational category (INSEE in 6 categories)
* Items of the ACR 1987 and ACR/EULAR 2010;
* Length of the RA
* Erosive or not (presence Yes / no)
* IgM rheumatoid factor (presence Yes / No)
* Anti CCP antbodies (presence Yes / No)

During follow-up visits (M3 and M6), the elements collected are:

1. by the study technician (TEC)

   * the inflammatory activity index, evaluated by patient (RAPID-3);
   * the functional limitations index (HAQ);
   * the PASS questionnaire;
   * the OM-RA-FLARE questionnaire;
   * the FLARE questionnaire.
2. by the doctor :

   * elements of DAS 28, this includes a blood test that will be done in the city or in the hospital ;
   * the doctor's decision at the end of the consultation, in terms of :

     * DMRADs: continuing the treatment, decreasing or increasing the dose, changing it due to its ineffectiveness, changing it due to patients' intolerance.
     * Symptomatic treatments: continuing corticosteroids, increase the dose of corticosteroids, corticosteroid infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Having Rheumatoid Arthritis (RA) since more than 6 months, meeting the ACR 1987 and the ACR / EULAR 2010;
* Treatment of RA:

  * Treatment of disease modifying anti-rheumatic drugs (DRMADs) or biological treatment stable for more than 2 months;
  * Symptomatic treatment (including corticosteroid) stable for more than 2 months;
* Receive the medical exam first;
* Agreed and signed the informed consent form;
* Ability to comply with the study protocol;
* Having the social insurance coverage

Exclusion Criteria:

* Patients undergoing surgery during the study period;
* Patients without any affiliation to a social security coverage (or entitled beneficiary);
* Patients under guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The validity of the questionnaire FLARE. | 6 mois
  The validity of the questionnaire shows the characteristics of the questionnaires (its ability to comprise the aspects for which it was designed). It will be studied by calculating the correlation coefficients between FLARE / OM-RA-FLARE on one hand, and various measures of disease activities (DAS 28, RAPID-3, RAID and AUC).

SECONDARY OUTCOMES:
The discriminating power of the instrument FLARE. | 6 mois.
  The discriminating power, i.e.the degree of precision for each particular instrument, considered individually, will be assessed by its reproducibility, sensitivity to change and its impact on medical decision making.
The feasibility of the questionnaire FLARE | 6 months.
  The feasibility will be measured by the percentage of non-calculable scores (missing data) and the number of items that are not filled for calculable scores.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PhD, Principal Investigator — CIC-EC Inserm, CHU de Nancy; Bruno Fautrel, MD, PhD, Principal Investigator — Service de Rhumatologie, Groupe Hospitalier Pitié - Salpêtrière, Paris; Jacques Morel, MD, PhD, Principal Investigator — Service d'immunorhumatologie, Hôpital Lapeyronie, Montpellier
Locations (13):
- France (13):
  - Service de Rhumatologie, CHU - Hôpital Sud A. Michallon, Grenoble, Auvergne-Rhône-Alpes
  - Service de Rhumatologie, CHU Hôpital Général, Dijon, Bourgogne-Franche-Comté
  - Service de Rhumatologie, CHU La Cavale Blanche, Brest, Brittany Region
  - Service de Rhumatologie, CHRU Hôtel Dieu, Nantes, Brittany Region
  - Service de Rhumatologie, CHU Jean Minjoz, Besançon, Franche-Comté
  - Service de Rhumatologie, CHU Fort de France, Fort de France, La Martinique
  - Service de Rhumatologie, Hôpitaux de Rouen, Rouen, Normandy
  - Service de Rhumatologie, APHP - CHU Bichat, Paris, Paris
  - Service de Rhumatologie, APHP - GH Pitié Salpêtrière, Paris, Paris
  - Service de Rhumatologie, CHU Conception, Marseille
  - Fédération de Rhumatologie, CHU Lapeyronie, Montpellier
  - Service de Rhumatologie, CHU de Poitiers, Poitiers
  - Service de Rhumatologie, Hôpital Larey, Toulouse

REFERENCES:
- [Derived] Fautrel B, Morel J, Berthelot JM, Constantin A, De Bandt M, Gaudin P, Maillefert JF, Meyer O, Pham T, Saraux A, Solau-Gervais E, Vittecoq O, Wendling D, Erpelding ML, Guillemin F; STPR Group of the French Society of Rheumatology. Validation of FLARE-RA, a Self-Administered Tool to Detect Recent or Current Rheumatoid Arthritis Flare. Arthritis Rheumatol. 2017 Feb;69(2):309-319. doi: 10.1002/art.39850. PMID 27636400